CLINICAL TRIAL: NCT06386263
Title: Real World Study of TrEatment Discontinuations and Modifications for Patients With HER2+ and HER2-low Metastatic Breast Cancer On Trastuzumab Deruxtecan
Brief Title: HER-TEMPO - Real World Treatment-related Outcomes on T-DXd in Canada
Acronym: HER-TEMPO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00032
Record Dates: First submitted 2024-04-03; First posted 2024-04-26 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Unresectable Breast Cancer; Metastatic Breast Cancer; HER2-low Expressing Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast Cancer; Metastatic breast cancer; HER-TEMPO; Trastuzumab Deruxtecan; Enhertu®; Observational
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HER2-positive: This cohort includes patients with HER2+ mBC who started treatment with T-DXd in the PSP.
  Interventions: Drug: Trastuzumab deruxtecan
- HER2-low: This cohort includes patients with HER2-low mBC who started treatment with T-DXd in the PSP.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — This is a non-interventional, observational study. Patients who are enrolled by their clinician will receive T-DXd per routine clinical practice through the PSP.
  Other Names: T-DXd; Enhertu

SUMMARY:
Trastuzumab deruxtecan (T-DXd) has been studied in multiple global prospective DESTINY-Breast trials and has a marketing authorization from Health Canada for patients with HER2-positive metastatic breast cancer (mBC) and HER2-low mBC, respectively.

Multiple stakeholders, including clinicians, patients, regulators, and healthcare decision makers, are interested in real-world treatment-related outcomes in order to better represent the effectiveness of therapies in routine care settings.

DETAILED DESCRIPTION:
This is a non-interventional, observational, hybrid (involving both primary and secondary data), cohort study that is utilizing patient support program (PSP) data. PSPs in Canada can support patients in accessing medicines after Health Canada has granted marketing authorization of a new drug or new indication before public reimbursement is available.

The outcomes will be assessed for the HER2-positive and HER2-low cohorts separately.

The primary objectives include assessing early treatment discontinuation rates at 3-, 6-, and 9-months after initiating T-DXd, and characterizing T-DXd dose modifications (i.e., interruptions and reductions) over the course of treatment for HER2+ mBC and HER2-low mBC.

Secondary objectives include estimating the real-world time to discontinuation (rwTTD) of T-DXd, reasons for treatment discontinuations, and real world duration of treatment and dose intensity with T-DXd.

The primary analysis population for all primary and secondary objectives will be the Total PSP Population (TPP), which includes all patients enrolled into the PSP who meet study criteria. Sensitivity analyses will also be performed in the Study PSP population (SPP), which will be a subset of patients from the TPP who provide study consent for additional data collection.

ELIGIBILITY:
Inclusion Criteria:

Enrollment criteria for HER2-positive PSP:

* Adults, 18 years of age or older
* Unresectable or metastatic HER2-positive breast cancer who have received at least one prior anti-HER2-based regimen either in the metastatic setting, or in the neoadjuvant or adjuvant setting and developed disease recurrence during or within 6 months of completing neoadjuvant or adjuvant therapy
* Patients must not have received a prior anti-HER2 ADC, such as trastuzumab emtansine, in the metastatic setting
* Patients who received a prior anti-HER2 ADC in the adjuvant setting must have progressed >12 months following the completion of therapy

Enrollment criteria for HER2-low PSP:

* Adults, 18 years of age or older
* Unresectable or metastatic HER2-low (IHC 1+ or IHC 2+/ISH-) breast cancer who have received at least one prior line of chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy
* Patients with HR+ breast cancer should have received at least one or be considered ineligible for endocrine therapy.

Patients in the SPP must additionally meet the following criteria:

* Patients must have provided consent to be contacted for future research and provided consent to participate in the current observational study

Exclusion Criteria (both cohorts):

* Patients who enrolled in the PSP, but did not initiate therapy with T-DXd by the end of the PSP program
* Patients with medical history of Interstitial Lung Disease (ILD) / pneumonitis that required steroids or current ILD /pneumonitis
* Patients who do not have adequate renal or hepatic function, defined as:
* Inadequate renal function is defined as Creatinine clearance <30 mL/min, as calculated using the Cockcroft-Gault equation .
* Inadequate hepatic function is aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >5 × upper limit of normal (ULN). Total bilirubin >1.5 × ULN if no liver metastases or ≥ 3 x ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable or metastatic HER2-positive or HER2-low breast cancer enrolled in the PSP who started treatment with T-DXd.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Early treatment discontinuation rates | 3, 6, 9 months
  Summary statistics of cumulative number and proportion of patients discontinuing at each timepoint
Dose modifications | from baseline to treatment discontinuation or the end of PSP, assessed up to 12 months (HER2-positive cohort) and up to 14 months (HER2-low cohort)
  Summary statistics about number and proportion of patients experiencing a dose modification (reduction or interruption) while receiving treatment in the PSP

SECONDARY OUTCOMES:
Real world time to treatment discontinuation (rwTTD) | from baseline to treatment discontinuation (self-report or recorded in the PSP database), end of the PSP, or end of the study period, assessed up to 24 months
  Median time from first dose of T-DXd to earliest date of T-DXd discontinuation as recorded in the patient support program (PSP) database or self-report from follow-up, or death, whichever occurs first
Reasons for treatment discontinuations | from baseline to treatment discontinuation (self-report or recorded in the PSP database), end of the PSP, or end of the study period, assessed up to 24 months
  Summary statistics about the number and proportion of patients with pre-specified reasons for treatment discontinuations as recorded by the clinician in the PSP program or based on self-report
Median treatment duration and dose intensity | from baseline to treatment discontinuation (as recorded in the PSP database) or end of the PSP, assessed up to 12 months (HER2-positive cohort) and up to 14 months (HER2-low cohort)
  Median treatment duration (and range, 95% CI): time from treatment initiation to treatment discontinuation excluding any dose interruptions; and dose intensity (DI) will be measured by the total drug delivered over the total time for the course of treatment (RDI will be the ratio of DI to the standard dose intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brezden-Masley, Principal Investigator — Sinai Health System
Locations (1):
- Research Site, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Brezden-Masley C, Qadeer R, Senhaji Mouhri Z, Salvo B, Bonar N, Spin P, Shokar S. Canadian real-world hybrid longitudinal cohort study of treatment discontinuations and modifications for patients with HER2+ and HER2-low metastatic breast cancer on trastuzumab deruxtecan enrolled in a patient support programme: the HER-TEMPO study protocol. BMJ Open. 2025 Sep 21;15(9):e100889. doi: 10.1136/bmjopen-2025-100889. PMID 40976668